CLINICAL TRIAL: NCT00927810
Title: A 24-week Open-label, Multicenter, Follow-up and Extension Study to CACZ885H2251, to Assess Safety, Tolerability and Efficacy of Canakinumab (ACZ885) in Patients With Gout Who Were Given Canakinumab at the Time of Gout Flare
Brief Title: Long Term Study of Canakinumab (ACZ885) in Patients With Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885H2251E1
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Gouty Arthritis
Keywords: Gouty; Gouty arthritis; Gout flares; Anti-interleukin-1β monoclonal antibody
MeSH Terms: conditions — Arthritis, Gouty | interventions — canakinumab

ARMS (1):
- canakinumab (Experimental)
  Interventions: Drug: Canakinumab

INTERVENTIONS:
Drug: Canakinumab

SUMMARY:
This 24-week open-label extension study is designed to provide additional long-term safety data up to a total of 1-year for patients rolling over from the core study, and to collect further efficacy and tolerability data for all the patients, irrespective whether they have an acute flare of gout or not. Patients will be treated on demand with canakinumab (ACZ885) in this extension study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the core study CACZ885H2251. A patient is defined as completing the core study if he/she completed the study up to and including the last visit (Visit 9).
* Patients who have signed a written informed consent before any trial procedure is performed.

Exclusion Criteria:

* Patients for whom continuation in the extension 1 is not considered appropriate by the treating physician.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive pregnancy test (serum or urine).
* Female patients who were physiologically capable of becoming pregnant, unless they were:

  * Female patients whose career, lifestyle, or sexual orientation precluded intercourse with a male partner.
  * Female patients whose partners had been sterilized by vasectomy or other means.
  * Using an acceptable method of contraception with a failure rate (Pearl Index (PI)) < 1.
  * Reliable contraception had to be maintained throughout the study and for 2 months after study drug discontinuation.

Other protocol defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2009-06-05 (Actual); Primary Completion 2010-08-04 (Actual); Study Completion 2010-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (42):
- Novartis Investigative site, Seattle, Washington, United States
- Novartis Investigative site, Capital Federal Buenos Aires, Argentina
- Novartis Investigative site, Jette, Belgium
- Colombia (4):
  - Novartis Investigative site, Barranquilla
  - Novartis Investigative site, Bogotá
  - Novartis Investigative site, Bucaramanga
  - Novartis Investigative site, Floridablanca
- Novartis Investigative site, Prague, Czech Republic, Czechia
- Germany (3):
  - Novartis Investigative site, Sachsen, Dresden / Schützenhöhe 16
  - Novartis Investigative site, Bayern, München / Mühlbaurstraße 16
  - Novartis Investigative site, Dessau, Roßlau / Kühnauer Straße 70 Sachsen- Anhalt
- Novartis Investigative site, Guatemala City, Guatemala
- Hungary (4):
  - Novartis Investigative site, Debrecen, Bartók B U 2-26
  - Novartis Investigative site, Kistarcsa, Semmelweis Tér 1.
  - Novartis Investigative site, Eger, Széchenyi U 27-29
  - Novartis Investigative site, Zalaegerszeg, Zrínyi U 1
- Poland (2):
  - Novartis Investigative site, Poznan
  - Novartis Investigative site, Wroclaw
- Novartis Investigative site, Lisbon, Portugal
- Russia (5):
  - Novartis Investigative site, Chelyabinsk
  - Novartis Investigative site, Moscow
  - Novartis Investigative site, Petrozavodsk
  - Novartis Investigative site, Saint Petersburg
  - Novartis Investigative site, Yaroslavl
- Novartis Investigative site, Singapore, Singapore
- Slovakia (5):
  - Novartis Investigative site, Bratislava
  - Novartis Investigative site, Košice
  - Novartis Investigative site, Nitra
  - Novartis Investigative site, Piešťany
  - Novartis Investigative site, Trenčín
- Novartis Investigative site, Pretoria, Gauteng, South Africa
- Novartis Investigative site, Madrid, Spain
- Taiwan (3):
  - Novartis Investigative site, Kaohsiung City
  - Novartis Investigative site, Taichung
  - Novartis Investigative site, Taipei
- Turkey (Türkiye) (6):
  - Novartis Investigative site, Ankara, Bahcellievler
  - Novartis Investigative site, Adana, Balcali
  - Novartis Investigative site, Izmir, Inciraltı
  - Novartis Investigative site, Aydin, Merkez
  - Novartis Investigative site, Manisa, Merkez
  - Novartis Investigative site, Gaziantep, Sehitkamil
- Novartis Investigative site, Jarrow, Tyne & Wear, United Kingdom

REFERENCES:
- [Result] Schlesinger N, Mysler E, Lin HY, De Meulemeester M, Rovensky J, Arulmani U, Balfour A, Krammer G, Sallstig P, So A. Canakinumab reduces the risk of acute gouty arthritis flares during initiation of allopurinol treatment: results of a double-blind, randomised study. Ann Rheum Dis. 2011 Jul;70(7):1264-71. doi: 10.1136/ard.2010.144063. Epub 2011 May 3. PMID 21540198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 75 centers in 18 countries.
Pre-assignment Details: A total of 341 participants enrolled in the study, out of which 330 participants completed the study.
Groups:
- Core: Canakinumab, Extension: 150 mg Canakinumab: Participants who were randomized to canakinumab in the core study (NCT00819585 [CACZ885H2251]), received single subcutaneous (SC) dose of 150 milligrams (mg) canakinumab (ACZ885) for at least one flare in this extension study (NCT00927810 [CACZ885H2251E1]).
- Core: Canakinumab, Extension: No Canakinumab: Participants who were randomized to canakinumab in the core study (NCT00819585 [CACZ885H2251]) and who did not received canakinumab in this extension study (NCT00927810 [CACZ885H2251E1]).
- Core: Colchicine, Extension: 150 mg Canakinumab: Participants who were randomized to colchicine in the core study (NCT00819585 [CACZ885H2251]), received single SC dose of 150 mg Canakinumab (ACZ885) for at least one flare in this extension study (NCT00927810 [CACZ885H2251E1]).
- Core: Colchicine, Extension: No Canakinumab: Participants who were randomized to colchicine in the core study (NCT00819585 [CACZ885H2251]) and who did not receive canakinumab in this extension study (NCT00927810 [CACZ885H2251E1]).
Period: Overall Study
Arm/Group | Core: Canakinumab, Extension: 150 mg Canakinumab | Core: Canakinumab, Extension: No Canakinumab | Core: Colchicine, Extension: 150 mg Canakinumab | Core: Colchicine, Extension: No Canakinumab
Started | 75 | 181 | 25 | 60
Completed | 75 | 173 | 24 | 58
Not Completed | 0 | 8 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 1
Not completed — Lost to Follow-up | 0 | 2 | 1 | 1
Not completed — Death | 0 | 2 | 0 | 0
Not completed — Abnormal laboratory value(s) | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Core: Colchicine, Extension: 150 mg Canakinumab: Participants who were randomized to colchicine in the core study (NCT00819585 [CACZ885H2251]), received single subcutaneous (SC) dose of 150 milligrams (mg) Canakinumab (ACZ885) for at least one flare in this extension study (NCT00927810 [CACZ885H2251E1]).
- Core: Colchicine, Extension: No Canakinumab: Participants who were randomized to colchicine in the core study (NCT00819585 [CACZ885H2251]) and who did not received canakinumab in this extension study (NCT00927810 [CACZ885H2251E1]).
- Total: Total of all reporting groups
Arm/Group | Core: Canakinumab, Extension: 150 mg Canakinumab | Core: Canakinumab, Extension: No Canakinumab | Core: Colchicine, Extension: 150 mg Canakinumab | Core: Colchicine, Extension: No Canakinumab | Total
Number analyzed (Participants) | 75 | 181 | 25 | 60 | 341
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (10.20) | 53.8 (11.39) | 52.0 (11.00) | 51.5 (9.45) | 52.6 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 13 | 0 | 7 | 22
  Male | 73 | 168 | 25 | 53 | 319
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 46 | 143 | 19 | 49 | 257
  Black | 2 | 6 | 1 | 1 | 10
  Asian | 11 | 10 | 2 | 2 | 25
  Native American | 1 | 3 | 0 | 1 | 5
  Pacific islander | 0 | 0 | 0 | 2 | 2
  Other | 15 | 19 | 3 | 5 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: Adverse events (AEs) were defined as any unfavourable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events (SAEs) were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalisation, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards
Time Frame: From start of study up to study completion (up to 14 months)
Population: Safety Set 1 consisted of all participants from the core study who entered the extension study.
Measure: Count of Participants; unit: Participants
Arm/Group | Core: Canakinumab, Extension: 150 mg Canakinumab | Core: Canakinumab, Extension: No Canakinumab | Core: Colchicine, Extension: 150 mg Canakinumab | Core: Colchicine, Extension: No Canakinumab
Number analyzed (Participants) | 75 | 181 | 25 | 60
Participants | 31 | 52 | 9 | 15

2. Secondary Outcome: Difference Change From Baseline in Participant's Gout Pain During First Flare
Description: Gout pain was assessed using Visual analogue scale (VAS) with a range of 0 to 100 where 0= no pain, 100= unbearable pain. Difference from time of study drug administration (pre-dose) was reported.
Time Frame: Baseline and Day 7
Population: Efficacy Set consisted of all participants who received at least one dose of canakinumab in this extension study (NCT00927810 [CACZ885H2251E1]. Here the number of participants analyzed signifies participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Core: Canakinumab, Extension: 150 mg Canakinumab | Core: Colchicine, Extension: 150 mg Canakinumab
Number analyzed (Participants) | 52 | 13
units on a scale | -51.7 (15.86) | -67.4 (21.69)

3. Secondary Outcome: Number of Participants Achieved Patient's Global Assessment of Response to Treatment (5-Point Likert Scale) Based on First, Second, Third Gout Flare Category
Description: Patient's global assessment of response to treatment is 5-point Likert scale:1.Excellent, 2.Good, 3.Acceptable, 4.Slight, 5.Poor. Lower the score better the outcome.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Core: Canakinumab, Extension: 150 mg Canakinumab | Core: Colchicine, Extension: 150 mg Canakinumab
Number analyzed (Participants) | 63 | 21
Participants
  1. Gout Flare: Excellent | 40 | 7
  1. Gout Flare: Good | 17 | 14
  1. Gout Flare: Acceptable | 5 | 0
  1. Gout Flare: Slight | 1 | 0
  1. Gout Flare: Poor | 0 | 0
  2. Gout Flare: Excellent: number analyzed (Participants) | 11 | 5
  2. Gout Flare: Excellent | 4 | 4
  2. Gout Flare: Good: number analyzed (Participants) | 11 | 5
  2. Gout Flare: Good | 6 | 1
  2. Gout Flare: Acceptable: number analyzed (Participants) | 11 | 5
  2. Gout Flare: Acceptable | 1 | 0
  2. Gout Flare: Slight: number analyzed (Participants) | 11 | 5
  2. Gout Flare: Slight | 0 | 0
  2. Gout Flare: Poor: number analyzed (Participants) | 11 | 5
  2. Gout Flare: Poor | 0 | 0
  3. Gout Flare: Excellent: number analyzed (Participants) | 3 | 1
  3. Gout Flare: Excellent | 2 | 0
  3. Gout Flare: Good: number analyzed (Participants) | 3 | 1
  3. Gout Flare: Good | 1 | 1
  3. Gout Flare: Acceptable: number analyzed (Participants) | 3 | 1
  3. Gout Flare: Acceptable | 0 | 0
  3. Gout Flare: Slight: number analyzed (Participants) | 3 | 1
  3. Gout Flare: Slight | 0 | 0
  3. Gout Flare: Poor: number analyzed (Participants) | 3 | 1
  3. Gout Flare: Poor | 0 | 0

4. Secondary Outcome: Number of Participants Achieved Physician's Global Assessment of Response to Treatment (5-Point Likert Scale) Based on First, Second, Third Gout Flare Category
Description: Physician's global assessment of response to treatment is 5-point Likert scale:1.Very good, 2.Good, 3.Fair, 4.Poor, 5.Very poor. Lower the score better the outcome.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Core: Canakinumab, Extension: 150 mg Canakinumab | Core: Colchicine, Extension: 150 mg Canakinumab
Number analyzed (Participants) | 69 | 23
Participants
  1. Gout Flare: Very Good | 37 | 13
  1. Gout Flare: Good | 28 | 10
  1. Gout Flare: Fair | 2 | 0
  1. Gout Flare: Poor | 2 | 0
  1. Gout Flare: Very Poor | 0 | 0
  2. Gout Flare: Very good: number analyzed (Participants) | 12 | 5
  2. Gout Flare: Very good | 5 | 3
  2. Gout Flare: Good: number analyzed (Participants) | 12 | 5
  2. Gout Flare: Good | 7 | 2
  2. Gout Flare: Fair: number analyzed (Participants) | 12 | 5
  2. Gout Flare: Fair | 0 | 0
  2. Gout Flare: Poor: number analyzed (Participants) | 12 | 5
  2. Gout Flare: Poor | 0 | 0
  2. Gout Flare: Very poor: number analyzed (Participants) | 12 | 5
  2. Gout Flare: Very poor | 0 | 0
  3. Gout Flare: Very Good: number analyzed (Participants) | 3 | 1
  3. Gout Flare: Very Good | 1 | 0
  3. Gout Flare: Good: number analyzed (Participants) | 3 | 1
  3. Gout Flare: Good | 2 | 1
  3. Gout Flare: Fair: number analyzed (Participants) | 3 | 1
  3. Gout Flare: Fair | 0 | 0
  3. Gout Flare: Poor: number analyzed (Participants) | 3 | 1
  3. Gout Flare: Poor | 0 | 0
  3. Gout Flare: Very poor: number analyzed (Participants) | 3 | 1
  3. Gout Flare: Very poor | 0 | 0

5. Secondary Outcome: Number of Participants Reported No Pain, No Swelling, Absent Erythema on Physician's Assessment of Tenderness, Swelling and Erythema in Most Affected Joint During the First Flare in Participants Treated With Canakinumab by Parameter, Visit and Group
Description: Tenderness was rated on a 0-3 point scale: 0="no pain", 1=patient states that "there is pain", 2=patient states "there is pain and winces", and 3=patient states "there is pain, winces and withdraws" on palpation or passive movement of the most affected joint. Swelling was rated on a 0-3 point scale: 0="no swelling", 1="palpable", 2="visible", and 3=bulging beyond the joint margins". Erythema was rated as present, absent, or not assessable. Assessments were performed at the flare and control visits.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Core: Canakinumab, Extension: 150 mg Canakinumab | Core: Colchicine, Extension: 150 mg Canakinumab
Number analyzed (Participants) | 69 | 24
Participants
  Tenderness-Flare Visit- No pain | 2 | 0
  Tenderness-Control Visit- No pain | 60 | 21
  Joint swelling-Flare Visit-No swelling | 5 | 0
  Joint swelling-Control Visit-No swelling | 61 | 22
  Erythema-Flare Visit-Absent | 21 | 4
  Erythema-Control Visit-Absent | 66 | 24

6. Secondary Outcome: Amount of Rescue Medication After Study Drug Intake in Participants Treated With Canakinumab by Flare Order, Medication and Group
Description: The amount of naproxen and prednisolone taken after receiving treatment for each of the first 3 flares was recorded.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Core: Canakinumab, Extension: 150 mg Canakinumab | Core: Colchicine, Extension: 150 mg Canakinumab
Number analyzed (Participants) | 68 | 24
milligrams (mg)
  1.Gout flare-Naproxen | 1086.8 (1592.72) | 954.6 (1130.19)
  1.Gout flare-Prednisolone | 4.6 (20.84) | 4.2 (20.41)
  2.Gout flare-Naproxen: number analyzed (Participants) | 12 | 5
  2.Gout flare-Naproxen | 650.0 (642.79) | 200.0 (447.21)
  2.Gout flare-Prednisolone: number analyzed (Participants) | 12 | 5
  2.Gout flare-Prednisolone | 1.3 (3.11) | 0.0 (0.00)
  3.Gout flare-Naproxen: number analyzed (Participants) | 4 | 1
  3.Gout flare-Naproxen | 250.0 (500.00) | 0.0 (0)
  3.Gout flare-Prednisolone: number analyzed (Participants) | 4 | 1
  3.Gout flare-Prednisolone | 0.0 (0.00) | 0.0 (0)

ADVERSE EVENTS:
Time Frame: From start of study up to study completion (up to 14 months)
Groups:
- Core: Canakinumab 25 mg: Participants received canakinumab 25 mg subcutaneously (sc) on Day 1; canakinumab placebo sc on Days 29, 57, and 85; and colchicine placebo orally once daily for 16 weeks.
- Core: Canakinumab 50 mg: Participants received canakinumab 50 mg sc on Day 1; canakinumab placebo sc on Days 29, 57, and 85; and colchicine placebo orally once daily for 16 weeks.
- Core: Canakinumab 100 mg: Participants received canakinumab 100 mg sc on Day 1; canakinumab placebo sc on Days 29, 57, and 85; and colchicine placebo orally once daily for 16 weeks.
- Core: Canakinumab 200 mg: Participants received canakinumab 200 mg sc on Day 1; canakinumab placebo sc on Days 29, 57, and 85; and colchicine placebo orally once daily for 16 weeks.
- Core: Canakinumab 300 mg: Participants received canakinumab 300 mg sc on Day 1; canakinumab placebo sc on Days 29, 57, and 85; and colchicine placebo orally once daily for 16 weeks.
- Core : Canakinumab Q4wk mg: Participants received canakinumab 50 mg sc on Days 1 and 29; canakinumab 25 mg sc on Days 57 and 85; and colchicine placebo orally once daily for 16 weeks.
- Core : Colchicine 0.5 mg: Participants received colchicine 0.5 mg orally once daily for 16 weeks and canakinumab placebo sc on Days 1, 29, 57, and 85.
Arm/Group | Core: Canakinumab 25 mg | Core: Canakinumab 50 mg | Core: Canakinumab 100 mg | Core: Canakinumab 200 mg | Core: Canakinumab 300 mg | Core : Canakinumab Q4wk mg | Core : Colchicine 0.5 mg | Core: Canakinumab, Extension: 150 mg Canakinumab | Core: Canakinumab, Extension: No Canakinumab | Core: Colchicine, Extension: 150 mg Canakinumab | Core: Colchicine, Extension: No Canakinumab
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/54 | 0/54 | 0/54 | 0/53 | 0/53 | 1/108 | 0/75 | 2/181 | 0/25 | 0/60
Serious Adverse Events (participants affected / at risk) | 2/55 | 2/54 | 3/54 | 3/54 | 3/53 | 1/53 | 6/108 | 4/75 | 6/181 | 0/25 | 1/60
Other Adverse Events (participants affected / at risk) | 21/55 | 15/54 | 14/54 | 14/54 | 15/53 | 14/53 | 21/108 | 21/75 | 19/181 | 6/25 | 4/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core: Canakinumab 25 mg (N=55) | Core: Canakinumab 50 mg (N=54) | Core: Canakinumab 100 mg (N=54) | Core: Canakinumab 200 mg (N=54) | Core: Canakinumab 300 mg (N=53) | Core : Canakinumab Q4wk mg (N=53) | Core : Colchicine 0.5 mg (N=108) | Core: Canakinumab, Extension: 150 mg Canakinumab (N=75) | Core: Canakinumab, Extension: No Canakinumab (N=181) | Core: Colchicine, Extension: 150 mg Canakinumab (N=25) | Core: Colchicine, Extension: No Canakinumab (N=60)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial fibrosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stupor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core: Canakinumab 25 mg (N=55) | Core: Canakinumab 50 mg (N=54) | Core: Canakinumab 100 mg (N=54) | Core: Canakinumab 200 mg (N=54) | Core: Canakinumab 300 mg (N=53) | Core : Canakinumab Q4wk mg (N=53) | Core : Colchicine 0.5 mg (N=108) | Core: Canakinumab, Extension: 150 mg Canakinumab (N=75) | Core: Canakinumab, Extension: No Canakinumab (N=181) | Core: Colchicine, Extension: 150 mg Canakinumab (N=25) | Core: Colchicine, Extension: No Canakinumab (N=60)
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2 | 3 | 1 | 0 | 2 | 2 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 2 | 2 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2 | 3 | 1 | 3 | 4 | 5 | 4 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 4 | 2 | 3 | 2 | 3 | 4 | 6 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 3 | 0 | 0 | 4 | 1 | 2 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 1 | 2 | 6 | 3 | 6 | 3 | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 4 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 6 | 2 | 2 | 5 | 4 | 2 | 1 | 6 | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.